CLINICAL TRIAL: NCT07200934
Title: Effect of Adding TENS to Mediterranean Diet on Appetite and Liver Enzymes in Nonalcoholic Fatty Liver Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Anwar Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005933
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Transcutaneous Electric Nerve Stimulation; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS + Mediterranean Diet (Experimental): This group will consist of 25 patients, who will receive TENS treatment at T6 dermatome for 30 minutes, 3 times per week for 12 weeks, in addition to following Mediterranean diet for 12 weeks.
  Interventions: Device: Transcutaneous electrical stimulation (TENS); Other: Mediterranean Diet
- Mediterranean Diet (Active Comparator): This group will consist of 25 patients, who will follow Mediterranean diet only for 12 weeks.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Device: Transcutaneous electrical stimulation (TENS) — The negative/active pad surface electrode will be applied at the T6 dermatome on the abdomen (is located at the left upper quadrant of the abdomen, 2 cm below the ribcage at the left midclavicular line) for stimulation and the passive/positive electrode will be applied on the left T6 costovertebral junction to complete the circuit.
  * The specific parameters of TENS will be burst mode, 2.0 Hz frequency, and 300 micro-seconds width
  * The patients will receive 3 times 30 min session each week for a period of consecutive 12 weeks.
  * The intensity of TENS will be gradually increased from 0 mA till the subject felt a comfortable tingling sensation beneath the electrode without any muscle contraction and pain.
  Arms: TENS + Mediterranean Diet
Other: Mediterranean Diet — The recommended composition of Mediterranean diet regimen: is characterized by a high intake of plant foods, fruits, vegetables, breads and other cereals (traditionally minimally refined), potatoes, beans, nuts and seeds; minimally processed, fresh fruits as a typical dessert, with sweets containing sugars or honey a few times per week; .a high intake of olive oil (especially virgin and extra-virgin olive oil) as the main source of fat; a moderate intake of dairy products (mostly as cheese and yoghurt); zero to four eggs per week; low to moderate amounts of fish and poultry; low amounts of red meat. The diet plan included generally 50% carbohydrates (from vegetables, fruits, legumes, and whole grains), 35% fats (from healthy oils, nuts, seeds, and fish), and 15% protein (from legumes, fish, nuts, dairy, poultry, and eggs).

SUMMARY:
This study aims to identify the effect of adding TENS to the Mediterranean diet on appetite and liver enzymes in Nonalcoholic fatty liver patients.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD), also termed metabolic dysfunction-associated fatty liver disease, is one of the most common chronic liver diseases worldwide. The development of NAFLD is fueled by a sedentary lifestyle, low frequency of physical activity, unhealthy diet and excessive calorie intake. NAFLD is characterized by fat accumulation in the liver accounting for >5% of hepatic tissue weight (fatty liver), as well as liver inflammation, which is not caused by alcohol abuse.

NAFLD prevalence is on the rise, mainly due to the presence of the obesity epidemic. Nowadays, NAFLD has been suggested to affect approximately 25% of the population worldwide. they have found a greater increase among men than women regarding the prevalence of NAFLD. Moreover, its mortality is projected to approach an increase of 65% to 100% by 2030 in Asian-Pacific regions.

Globally, NAFLD prevalence averages 24.1%, ranging from 13.5% in Africa to 31.8% in the Middle East. Despite limited data on the extent of NAFLD in Egypt, the available data indicate a prevalence of nearly 32% among Egyptians, compared to a global prevalence of 25% Egypt ranks among the top ten countries with the highest obesity rates in the world.

Lifestyle modifications are the cornerstone of NAFLD management. A Mediterranean diet (MD), rich in whole grains, vegetables, fruits, nuts, and olive oil, is proven to improve liver health by reducing inflammation and fat accumulation.

Transcutaneous electrical stimulation (TENS) of T6 dermatome on the abdomen generates impulses which are carried to the spinal cord via afferent pathways, in turn, efferent impulses pass through the vagus nerve, and effects are induced similar to the gastric stimulator .This somato-autonomic reflex helps in decreasing appetite.

Therefore, the primary aim of this study it will impact future researcher about the beneficial effect of T6 dermatomal stimulation by the transcutaneous method in managing obesity, improving liver function and finally promoting body health related measure in non-alcoholic fatty liver patients.

ELIGIBILITY:
Inclusion Criteria:

* The age will range from 35-45 years old.
* BMI (Body Mass Index 30-34.9 kg/m2.)
* With fatty liver infiltration confirmed by abdominal ultrasound
* Elevated of liver enzymes as a primary marker
* All patients are psychologically stable.

Exclusion Criteria:

* History of cardiovascular or respiratory disease.
* If any known endocrine diseases e.g. Hypothyroidism (which elevates liver enzymes and effects on appetite)
* Any acute or chronic illness causing elevated liver enzymes other than fatty liver e.g. Hepatitis b, Hepatitis c
* Any neurological illness or impairment can effect on sensation
* Patients associated with infections, mental or malignant conditions.
* Patients who have undergone any gastric surgery e.g. Bariatric surgery
* Taking dietary supplement for weight reduction.
* Patients who participating in any other exercise program.

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale for appetite (VAS) | 12 weeks
  This method is used to evaluate the appetite level of fatty liver patients before and after treatment procedures. This method usually consists of a set of questions assessing hunger, fullness/satisfaction, desire to eat and prospective food intake the question is presented with a 100 mm horizontal line scale.
Levels of liver transaminases aspartate transaminase (AST) | 12 weeks
  It will be measured pre and post-treatment for all participants in both groups.
Levels of liver alanine transaminase (ALT) | 12 weeks
  It will be measured pre and post-treatment for all participants in both groups.

SECONDARY OUTCOMES:
Body mass index (BMI) | 12 weeks
  The BMI will be measured before and after treatment to measure the success of treatment procedures in losing weight for fatty liver patients.
Relative fat mass (RFM) | 12 weeks
  The ratio of the patient's height and waist measurement, both in meters, is multiplied by 20 before being subtracted from a number that adjusts for differences in gender and height: RFM for adult Males: 64 - 20 × (height / waist circumference).This method is used to measure the success of treatment procedures in reducing fat mass of fatty liver patients.
Fatigue Severity Scale (FSS) | 12 weeks
  Fatigue is considered the most common symptom for fatty liver patients Therefore we use this scale before and after treatment procedures. The FSS is a nine-item, self-reported questionnaire. Each item includes a seven-point, Likert-type response where 1 = "strongly disagree" and 7 = "strongly agree." indicates strong agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen Ghareeb El-Nahas, PhD, Study Chair — Professor, Cairo university; Salma Ibrahim AL Ghitany, PhD, Study Director — Lecturer, Cairo university; Shawky Abdelhamid Fouad Abdel Gawad, Study Director — Professor, Cairo university
Locations (1):
- Internal Medicine Hospital Cairo University, Giza, Egypt